CLINICAL TRIAL: NCT03977636
Title: Determinants of Time Required by Medical Information Technicians for Quality Control of Hospital Activity Coding, in French Medico-administrative System
Brief Title: Determinants of Time Required by Medical Information Technicians for Quality Control of Hospital Activity Coding
Acronym: DALDIM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-09Obs-CHRMT
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Quality Control
Keywords: Diagnosis-related groups; Activity-based funding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since 2008, in France, hospital funding is determined by the nature of activities provided (activity-based funding). Quality control of hospital activity coding is essential to optimize hospital remuneration. There is a need for reliable tools to allocate human resources wisely in order to improve these controls.

DETAILED DESCRIPTION:
The main objective of this study was to identify the determinants of time needed by medical information technicians to control hospital activity coding in a Regional Hospital Center.

From March 2016 to the beginning of January 2017, medical information technicians reported the time they spent on each quality control, and the time they needed when they had to code the entire stay. Multiple linear regressions were performed to identify the determinants of quality control or coding duration. A split sample validation was used: model was created on one half of the sample and validated on the remaining half.

ELIGIBILITY:
Inclusion Criteria:

* To be admitted to a medical unit of the CHR Metz Thionville

Exclusion Criteria:

* Any exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the Regional Hospital of Metz-Thionville
Sampling Method: Non-Probability Sample
Enrollment: 5431 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Time for quality control | Day 1
  medical information technicians reported the time they spent on each quality control

SECONDARY OUTCOMES:
Time to code the entire stay | Day 1
  medical information technicians reported the time they needed when they had to code the entire stay